CLINICAL TRIAL: NCT00296855
Title: Intra-individual Open-label Multicenter Comparison Study of Magnetic Resonance Angiography (MRA) With the Blood Pool Contrast Agent Vasovist® and a Conventional Extracellular Contrast Agent With Intra-arterial Digital Subtraction Angiography (i.a. DSA) in Patients With Peripheral Artery Disease
Brief Title: Comparison Study of Vasovist® Magnetic Resonance Angiography (MRA) and an MRA With a Conventional Extracellular Contrast Agent With X-ray Angiography in Patients With Peripheral Artery Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91463; EudraCT No. 2005-002547-66; 308861
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral artery disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease | interventions — gadofosveset trisodium

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Vasovist (BAY86-5283, MS-325)

INTERVENTIONS:
Drug: Vasovist (BAY86-5283, MS-325) — All patients receive a single IV bolus injection of Vasovist at a dose of 0,03 mmol/kg BW at a flowrate of 0,5 mL/sec, followed by a saline flush of at least 30 mL

SUMMARY:
The particular aim of this study is the comparison of the diagnostic results of MRA images upon application of Vasovist (gadofosveset), a contrast agent not yet available on the market, with the MRA images upon application of a conventional extracellular contrast agent. A catheter angiography, which will be performed as a routine diagnostic procedure for vascular diseases, will serve as an evaluation standard.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a certain circulation disorder (aortoiliac disease Fontaine-stage IIb / IV) and an indication for the evaluation of the peripheral run-off arteries from the infrarenal aorta to the calves
* Patients who are scheduled for X-ray angiography and magnetic resonance angiography (MRA) of the arteries mentioned above
* Patients who have had a contrast-enhanced MRA examination of the arteries mentioned above using a standard extracellular contrast agent performed within 1 - 7 days prior to the study MRA examination

Exclusion Criteria:

* Less than 18 years of age
* Women who are pregnant, breast feeding or who are of childbearing potential and have not had a negative urine pregnancy test the same day as the study MRA examination
* Requiring immediate therapy for their vascular disease or in whom conduct of all three angiographic procedures is not possible
* Not being able to remain lying down for at least 45 - 60 min
* Patients with a history of serious allergic reactions to any allergen including drugs and contrast agents or with a history of sickle cell disease or other hemolytic anemia
* Having any contraindication to magnetic resonance imaging (MRI) examination or specifically for MRA (e.g. pacemaker, recent wound clips, and severe claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2006-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic potential of Vasovist enhanced MRA | Imaging after baseline visit, before and after Vasovist injection

SECONDARY OUTCOMES:
Comparison of the quantitative assessment and the qualitative assessment of arterial stenosis/disease as compared to X-ray angiography | After imaging
Quantitative assessment of vessel enhancement | After imaging
Qualitative assessment of disease | After imaging
Qualitative assessment of plaque morphology | After imaging
Evaluation of quality of vascular anatomy and delineation of vessel wall, venous enhancement and diagnostic potential of venous enhancement | After imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (22):
- Argentina (3):
  - Buenos Aires, Buenos Aires
  - Lornas de Zamora, Buenos Aires
  - Buenos Aires, Buenos Aires F.D.
- Austria (3):
  - Sankt Pölten, Lower Austria
  - Graz, Styria
  - Vienna, Vienna
- Brazil (3):
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - São Paulo, São Paulo
- Germany (8):
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Berlin, State of Berlin
- Mexico (3):
  - Monterrey, Nuevo León
  - Mexico D. F.
  - México D.F.
- Switzerland (2):
  - Basel, Basel
  - Baden